CLINICAL TRIAL: NCT05985005
Title: The Effectiveness of a Chatbot-facilitated High Alert Medication Education for 2-year Post Graduate Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20221007R
Record Dates: First submitted 2023-05-23; First posted 2023-08-09 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-05

CONDITIONS: Education, Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online simulation of high alert medication safety training (Experimental)
  Interventions: Other: online simulation of high alert medication safety training
- classroom teaching regarding high alert medication (No Intervention)

INTERVENTIONS:
Other: online simulation of high alert medication safety training — online simulation of high alert medication safety training
  Arms: online simulation of high alert medication safety training

SUMMARY:
This study involves three stages. In the first stage, qualitative research design is used to understand clinical nurses' learning needs on high alert medication. In the second stage, " high alert medication knowledge inventory " and " high alert medication safety inventory " will be developed based on the literature and results from qualitative study in the stage one. In the third stage, randomized control trail study design will be used. The nursing staffs in the experimental group receive " online simulation of high alert medication safety training ", the staffs from the control group receive classroom teaching regarding high alert medication". A total of 124 nurses will be invited to participate in this study, 62 subjects will be assigned in each group . After the intervention, we will examine the learning effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Nursing staff who are licensed and have passed the Medication Safety Course for Newcomers to independently perform drug delivery techniques.
2. Nursing staff who are willing to participate in this research and complete the research consent form.

Exclusion Criteria:

1. Not fully involved in the study
2. Nursing staff not involved in dispensing medicine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
high alert medication knowledge inventory | Change from Baseline high alert medication knowledge inventory at 1 months
  Nurse ' medication knowledge
high alert medication safety inventory | Change from high alert medication safety inventory at 1 months
  Nurse ' medication safety
Learning Engagement Scale | Change from high alert medication safety inventory at 1 months
  Nurse ' Learning Engagement Scale

SECONDARY OUTCOMES:
Learning satisfaction | through study completion, an average of 1 Week
  Learning satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- He Ting-I, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol
Time Frame: starting in January 2025 until January 2030